CLINICAL TRIAL: NCT05835622
Title: Clinical Investigation of the Quality of Life Benefit of Using a Home Walking Exoskeleton for a Population of Multiple Sclerosis Patients With Gait Disorders.
Brief Title: Clinical Investigation of the Quality of Life Benefit of Using a Home Walking Exoskeleton for a Population of Multiple Sclerosis Patients.
Acronym: EXHOMESEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pôle Saint Hélier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-A03094-37
Record Dates: First submitted 2023-04-04; First posted 2023-04-28 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: After screening visit, patients are randomised between two Arms. Patients in Arm A start with experimental phase and after a wash-out period start the control phase (without exoskeleton). Patients randomised in Arm B start with the control phase and after the wash-out period start the experimental phase. After that, all patients have a follow-up period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Other): 8 weeks of using keeogo at home (experimental phase) followed by 8 weeks of wash-up and then followed by 8 weeks of recommended home practise (control phase).
  Interventions: Device: Keeogo; Other: adviced home practice
- Arm B (Other): 8 weeks of recommended home practise (control phase) followed by 8 weeks of wash-up and then followed by 8 weeks of using keeogo at home (experimental phase)
  Interventions: Device: Keeogo; Other: adviced home practice

INTERVENTIONS:
Device: Keeogo — Keeogo is exoskeleton for walking assistance
Other: adviced home practice — health tips for regular and appropriate physical activity

SUMMARY:
The goal of this clinical investigation is to evaluate the effectiveness of home use of a lightweight robotic lower limb exoskeleton as a walking aid device on quality of life in patients with multiple sclerosis with gait disorders.

Participants will wear an exoskeleton (Keeogo) for 8 weeks at home during the experimental phase. This phase is compared to an 8-week control phase at home with advice on regular physical activity adapted to their abilities.

DETAILED DESCRIPTION:
It is a multicenter, controlled, randomized, cross-over, open-label clinical investigation.

Patients with multiple sclerosis with an Expanded Disability Status Scale (EDSS) between 5 and 6.5,living at home and using an assistive device for walking will be included.

After enrollment, patients will be randomised in one of the 2 study-arm.

* Arm A: experimental phase / Wash-Out (WO) (8 weeks) / control phase
* Arm B: control phase / WO (8 weeks) / experimental phase

During the experimental phase, patients will receive a Keeogo specific training for five days. The purpose of this training programme is to ensure familiarity and acceptance of the device. Then, the patients will take Keeogo home and will have to use the device as much as possible indoors and outdoors for seven weeks.

During the control phase, patients will be at home for eight weeks with advice on regular physical activity adapted to their abilities.

After the second phase, all patients will have a 3 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient with multiple sclerosis according to the revised Mac Donald diagnostic criteria (2017) in the relapsing-remitting form more than 6 months from a relapsing or progressive period.
* An Expanded Disability Status Scale (EDSS) between 5 and 6.5 on the EDSS scale (Kurtzke 1983)
* Living at home
* Using a walking aid
* 18 years old or older
* Have freely consented to participate in this study
* To be more than 1m52 tall
* Hip Manual Muscle Testing (MMT) score ≥ 3+ (flexors and expanders)
* Knee Manual Muscle Testing (MMT) score ≥ 2 (flexors and expanders)
* Berg scale (BBS) score > 20
* Patient affiliated with a social security plan or beneficiary of such a plan.

Non-Inclusion Criteria:

* Impaired comprehension preventing completion of the protocol
* Inability to walk without assistance for 10 minutes
* Have a rehabilitation stay scheduled during the follow-up period of the clinical investigation
* Diagnosed psychiatric conditions that may have an impact on the experience of withdrawal of technical assistance at the end of the protocol
* Severe cognitive impairment (MMSE<24)
* Person deprived of liberty by a judicial or administrative decision
* A person under psychiatric care or admitted to a health or social institution for purposes other than research.
* Spasticity >3 on the Held and Tardieu scale affecting the hamstring, quadriceps, adductor or sural triceps muscles
* Complete paralysis of the lower limbs
* Severe osteoporosis
* Hip and/or knee replacements that would sufficiently limit range of motion for walking and sitting or squatting
* Severe vascular disorders of the lower limbs
* Existing wounds or skin lesions where the device is worn
* Pregnant woman or postpartum woman who has not completed lumbopelvic recovery
* Orthopedic disorders of the lower limb that may prevent satisfactory adjustment of Keeogo
* Uncontrolled epilepsy or tremors
* Uncontrolled autonomic dysreflexia
* Severe balance disorders, neurological disorders (any condition that prevents the safe control of balance and/or movement of the limbs at all times while wearing the Keeogo System)
* Conditions that prevent safe moderate-intensity exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
Evolution of the quality of life assessed with the "Functional Assessment Of Multiple Sclerosis" questionnaire (change between two time points) | Screening visit and visit after experimental phase (Week 8 for Arm A; Week 24 for Arm B)
  The Functional Assessment Of Multiple Sclerosis (FAMS) is a self-administered health questionnaire related to quality of life for patients with multiple sclerosis

SECONDARY OUTCOMES:
Walking and balancing performance with the Keeogo exoskeleton (1) | after experimental phase (Week 8 for Arm A; Week 24 for Arm B)
  Measured by 2 minutes walking test
Walking and balancing performance with the Keeogo exoskeleton (2) | after experimental phase (Week 8 for Arm A; Week 24 for Arm B)
  Measured by 10 meter walking test
Walking and balancing performance with the Keeogo exoskeleton (3) | after experimental phase (Week 8 for Arm A; Week 24 for Arm B)
  Measured by the Timed up and go Test
Walking and balancing performance with the Keeogo exoskeleton (4) | after experimental phase (Week 8 for Arm A; Week 24 for Arm B)
  Measured by Functional Stair Test (FST)
Walking and balancing performance with the Keeogo exoskeleton (5) | after experimental phase (Week 8 for Arm A; Week 24 for Arm B)
  Measured by the Sit to Stand Test (SST)
Walking and balancing performance with the Keeogo exoskeleton (6) | after experimental phase (Week 8 for Arm A; Week 24 for Arm B)
  Evaluations of spatio-temporal gait parameters using an instrumented walking system (Gaitrite®, Vicon® or Locometer® for example)
Spasticity of the quadriceps, hamstrings and abductors muscles | At all study visits (Screening, Week 8, Week 16, Week 24, Month 9)
  Assessed manually by the Held and Tardieu Test
Sense of self-efficacy | At all study visits (Screening, Week 8, Week 16, Week 24, Month 9)
  Measured by the Rosenberg Self-Efficacy Questionnaire
The average daily distance travelled | At study visits (Week 8, Week 24, Month 9)
  Measured by inertial units tracing the daily activity of the participants (descriptive daily distance travelled)
Fatigue | At all study visits (Screening, Week 8, Week 16, Week 24, Month 9)
  Measured by the French version of the fatigue impact scale in multiple sclerosis (EMIF-SEP) scored from 0 to 100% a low score is a better outcome
Anxiety and depression | At all study visits (Screening, Week 8, Week 16, Week 24, Month 9)
  Measured by the Hospital Anxiety and Depression score (HAD) scored from 0 to 21 for both subtitles (Anxiety and depression) a low score is a better outcome
Satisfaction with this new home technical aid | After experimental phase (Week 8 for Arm A; Week 24 for Arm B)
  Evaluated via the French version of the QUEST questionnaire (ESAT questionnaire)
Projection in use | After experimental phase (Week 8 for Arm A; Week 24 for Arm B)
  Evaluated by a usage questionnaire (UTAUT-based already used in a walking exoskeleton context)
Walking and balancing performance without exoskeleton (1) | At all study visits (Screening, Week 8, Week 16, Week 24, Month 9)
  Measured by the 2 minutes walking test
Walking and balancing performance without exoskeleton (2) | At all study visits (Screening, Week 8, Week 16, Week 24, Month 9)
  Measured by the 10 meter walking test
Walking and balancing performance without exoskeleton (3) | At all study visits (Screening, Week 8, Week 16, Week 24, Month 9)
  Measured by the Timed up and go Test
Walking and balancing performance without exoskeleton (4) | At all study visits (Screening, Week 8, Week 16, Week 24, Month 9)
  Measured by the Functional Stair Test (FST)
Walking and balancing performance without exoskeleton (5) | At all study visits (Screening, Week 8, Week 16, Week 24, Month 9)
  Measured by the Sit to Stand Test (SST)
Walking and balancing performance without exoskeleton (6) | At all study visits (Screening, Week 8, Week 16, Week 24, Month 9)
  Evaluations of spatio-temporal gait parameters using an instrumented walking system (Gaitrite®, Vicon® or Locometer® for example)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gallien, Doctor, Principal Investigator — Pole Saint-Hélier
Locations (6):
- France (6):
  - Hospices Civils de Lyon - Hôpital Henry Gabrielle, Saint-Genis-Laval, Auvergne-Rhône-Alpes
  - Pôle Saint Hélier, Rennes, Brittany Region
  - Hôpital Saint Philibert-Groupement des Hôpitaux de l'Institut Catholique de Lille, Lomme, Hauts-de-France
  - Centre de rééducation Fonctionnelle Propara-Montpellier, Montpellier, Occitanie
  - CHU Angers- SSR Les Capucins, Angers, Pays de la Loire Region
  - CHU Nantes site de Saint Jacques, Nantes, Pays de la Loire Region

IPD SHARING:
Plan to Share IPD: No